

| Serial number |
|---------------|

## **Consent Form**

Title: The development of intracranial pressure control strategy and CSF neuro-biomarkers as neurologic prognostic factors in cardiac arrest patients treated with target temperature management

- 1. I understand an explanation of the clinical study, read the study descriptions, and discussed the study with the researchers satisfactorily.
- 2. I have heard about the risks and benefits of the study and have answered my questions satisfactorily.
- 3. I voluntarily agree to participate in this study.
- 4. I understand that I can refuse to participate in the study or withdraw participation in the study at any time without affecting future treatment, and I know that this decision will not harm me.
- 5. By signing this manual and consent, I agree that my personal information will be collected and processed by the researcher for the purposes of medical research to the extent permitted by current laws and regulations.
- 6. I understand that I will have a copy of the study description and consent form.

| Name of Participant | Sign | Date(Day/Mon/Year) |
|---------------------------|--------------------|--------------------|
| Name of Researcher | Sign | Date(Day/Mon/Year) |
| Name of Research Director | Sign | Date(Day/Mon/Year) |
| Legal Representative Name | Sign | Date(Day/Mon/Year) |
| Relationship | Reason for consent | |

NCT number: not yet assigned 25 October 2019